CLINICAL TRIAL: NCT05497141
Title: Dawneo Neoblazar® Transcatheter Tricuspid Valve Edge-to Edge Repair System Pivotal Clinical Trial (NoTR): A Trial to Evaluate the Safety and Effectiveness of Transcatheter Valve Edge-to-edge Repair System in Patients With Severe Tricuspid Regurgitation
Brief Title: Dawneo Neoblazar® Transcatheter Tricuspid Valve Edge-to Edge Repair System Pivotal Clinical Trial in Patients With Severe Tricuspid Regurgitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022YLK17
Record Dates: First submitted 2022-08-07; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Tricuspid Regurgitation
Keywords: sever tricuspid regurgitation; edge-to edge repair system; heart failure
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tricuspid valve edge-to edge Repair group (Experimental): Subjects who received Neoblazar® Transcatheter Tricuspid Valve Edge-to Edge Repair System will be included in this arm
  Interventions: Device: Neoblazar® Transcatheter Tricuspid Valve Edge-to Edge Repair System

INTERVENTIONS:
Device: Neoblazar® Transcatheter Tricuspid Valve Edge-to Edge Repair System — Subjects who received Neoblazar® Transcatheter Tricuspid Valve Edge-to Edge Repair System will be included in this arm. The Neoblazar® is intended for reconstruction of the insufficient tricuspid valve through tissue tissue approximation.

SUMMARY:
To evaluate the safety and effectiveness of Dawneo Neoblazar® transcatheter tricuspid valve edge-to-edge repair system in patients with severe tricuspid regurgitation.

This is a prospective, multicenter, randomized, objective performance criteria trial. 98 patients who meet the inclusion criteria will be included in the study. This study will be conducted in in each site as run-in subjects. Subjects who meet the requirements and who voluntarily participate in the trial and sign the informed consent form, will be implanted with the Neoblazar® Transcatheter Tricuspid Valve Edge-to Edge Repair System.

DETAILED DESCRIPTION:
OBJECTIVES：To evaluate the safety and effectiveness of Dawneo Neoblazar® transcatheter tricuspid valve edge-to-edge repair system in patients with severe tricuspid regurgitation.

CLINICAL INVESTIGATION POPULATION:Patients who are on echocardiographic evidence of severe tricuspid regurgitation.

CLINICAL INVESTIGATION DESIGN:This is a prospective, multicenter, single arm, objective performance criteria trial. 98 patients who meet the inclusion criteria will be included in the study. This study will be conducted in in each site as run-in subjects. Subjects who meet the requirements and who voluntarily participate in the trial and sign the informed consent form, will be implanted with the Neoblazar® Transcatheter Tricuspid Valve Edge-to Edge Repair System.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of age > 18 years;
2. Subjects suffering from severe tricuspid regurgitation (TR≥3+), defined by TTE or TEE;
3. Subject has symptoms with NYHA ≥ Class II-Iva, or at least one hospitalization for symptoms of heart failure during the past 12 months.
4. Subjects with two cardiac surgeons agreements of contraindications to surgery or high risk, who meets at least one of the following three conditions:

   ① Euroscore≥8%；

   ② Presence of 2 or more Frailty Index；

   ③ Presence of 2 or more organ insufficiencies。
5. Subjects who's tricuspid valve anatomy are suitable for transcatheter valve edge-to-edge repairment as assessed.
6. Subjects agreeing to the scheduled follow up requirements, who can understand the purpose of the clinical investigation, and sign voluntarily the informed consent form by themselves and/or the subject' legal guardians.

Exclusion Criteria:

1. Pulmonary artery systolic pressure >70 mmHg measured by transthoracic echocardiography or right heart catheterization, or irreversible precapillary pulmonary hypertension;
2. The presence of calcification in the grasping area of the tricuspid valve leaflets (including the anterior, septal, and posterior leaflets) that affects clamping, and the thickness of the tricuspid valve leaflets≥4mm;
3. Severe tricuspid leaflet perforation, cleft or other lesions which preventing the implantation;
4. Tricuspid valve leaflets coaptation gap >7mm
5. Tricuspid stenosis as assessed by echocardiography (defined as tricuspid orifice area ≤1.0 cm2)
6. LVEF≤20%；
7. Refractory heart failure requiring advanced intervention (e.g., left ventricular assist device, heart transplantation, etc.) (ACC/AHA stage D heart failure);
8. Myocardial infarction or unstable angina within 4 weeks;
9. Untreated severe coronary artery stenosis requiring revascularization;
10. Received percutaneous coronary intervention within 1 month prior to implantation;
11. Severe and uncontrolled hypertension: SBP≥180mmHg or DBP≥110mmHg;
12. Previously implantation of tricuspid valve, annuloplasty ring or accepted tricuspid valve repair surgery;
13. Pacemaker leads or ICD leads that may affect implantation
14. Complications of other cardiac diseases requiring surgical intervention;
15. Tricuspid leaflet lesions due to rheumatic heart disease (e.g., leaflet grossness, thickening, poor compliance, etc.);
16. Combined with moderate or severer aortic stenosis, aortic regurgitation, mitral stenosis, mitral regurgitation;
17. Congenital Ebstein malformation;
18. Presents of thrombus, vegetation, mass in the right heart system, femoral vein or inferior vena cava, etc.
19. Hemorrhagic disease or hypercoagulable state;
20. Contraindication or allergic reaction to dual antiplatelet agents and anticoagulants;
21. Active infection requiring antibiotic treatment;
22. Renal failure, requiring dialysis treatment;
23. Severe terminal illness (e.g., cancer, etc.) with a life expectancy of less than 1 year;
24. Pregnant, lactating women, women preparing to conceive or women of childbearing age with a positive HCG test (except for women whose medical history describes menopause);
25. Subjects have not met the observed endpoint in other clinical studies in which they participated;
26. Inability to comply with the clinical investigation follow-up or other clinical investigation requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-08-22 (Estimated); Study Completion 2023-10-22 (Estimated)

PRIMARY OUTCOMES:
Rate of Implantation Success | 12 months
  1. No all-cause mortality after implantation;
  2. No tricuspid open surgery after implantation;
  3. tricuspid regurgitation reduction at least 1 grade.

SECONDARY OUTCOMES:
Initial Success | 1 week
  The device was successfully delivered to the target position and successfully released, and the delivery system was successfully withdrawn from the body without any detachment incident.
NYHA Functional Class | 30 days, 6 months, 12 months, annual for five years
  New York Heart Association functional class（NYHA). Number of Improvement in NYHA classification is defined as a reduction in NYHA classification of at least 1 grade from baseline by Core Lab assessment.
Six-minute walk test | 30 days, 6 months, 12 months, annual for five years
  Change in distence(m) from baseline
Reduction in TR grade | 30 days, 6 months, 12 months, annual for five years
  Number of patients with reduction in TR from baseline by Core Lab assessment

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Dr, Principal Investigator — Clinical Trial Center of Xiamen Cardiovascular Hospital; Nianguo Dong, Dr, Principal Investigator — Wuhan Xiehe Hospital
Locations (1):
- Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian, China